CLINICAL TRIAL: NCT03545191
Title: Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group, Polysomnography Study to Assess the Efficacy and Safety of ACT-541468 in Adult and Elderly Subjects With Insomnia Disorder
Brief Title: Study to Assess the Efficacy and Safety of ACT-541468 (Daridorexant) in Adult and Elderly Subjects With Insomnia Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-078A301
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Results first posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — daridorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Daridorexant 25 mg (Experimental)
  Interventions: Drug: Daridorexant 25 mg
- Daridorexant 50 mg (Experimental)
  Interventions: Drug: Daridorexant 50 mg
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Daridorexant 25 mg — Daridorexant will be administered as tablets, orally, once daily in the evening.
  Arms: Daridorexant 25 mg
Drug: Daridorexant 50 mg — Daridorexant will be administered as tablets, orally, once daily in the evening.
  Arms: Daridorexant 50 mg
Other: Placebo — Matching placebo will be administered as tablets, orally, once daily in the evening.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess efficacy and safety of ACT-541468 (daridorexant) in adult and elderly subjects with insomnia disorder. Efficacy will be evaluated on objective and subjective sleep parameters.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure;
* Male or female aged ≥ 18 years;
* Insomnia disorder according to DSM-5 criteria;
* Insomnia Severity Index score ≥ 15;
* Insufficient sleep quantity as collected subjectively in the sleep diary;
* Women of childbearing potential must have a negative and urine pregnancy test and use the contraception scheme up to at least 30 days after last study treatment intake.

Exclusion Criteria:

* Body mass index below 18.5 or above 40.0 kg/m2;
* Any lifetime history of of related breathing disorder, periodic limb movement disorder, restless legs syndrome, circadian rhythm disorder, rapid eye movement (REM) behavior disorder, narcolepsy, or apnea/ hypopnea;
* Cognitive behavioral therapy (CBT) only allowed if, the treatment started at least 1 month prior to Visit 3 and the subject agrees to continue this CBT throughout the study;
* Self-reported usual daytime napping ≥ 1 hour per day and ≥ 3 days per week;
* Acute or unstable psychiatric conditions diagnosed by the Mini International Neuropsychiatric Interview;
* Mini Mental State Examination (MMSE) score < 25 in subjects ≥ 50 years;
* For female subjects: pregnant, lactating or planning to become pregnant during projected duration of the study;
* History or clinical evidence of any disease or medical condition or treatment, which may put the subject at risk of participation in the study or may interfere with the study assessments.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 930 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-01-25 (Actual); Study Completion 2020-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (81):
- United States (36):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Pulmonary Associates of the Southeast/WCR, Birmingham, Alabama
  - Preferred Research Partners, Inc, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - Marvel Clinical Research, Huntington Beach, California
  - Long Beach Clinical Trials, Long Beach, California
  - Artemis Institute for Clinical Research, San Diego, California
  - PAB Clinical Research, Brandon, Florida
  - St. Francis Sleep Allergy and Lung Institute, Clearwater, Florida
  - Innovative Clinical Research, Inc., Hialeah, Florida
  - Research Centers of America, Hollywood, Florida
  - Canvas Clinical Research, LLC, Lake Worth, Florida
  - BioMed Research Institute, Miami, Florida
  - Clinical Site Partners, LLC, Winter Park, Florida
  - LaPorte County Institute for Clinical Research, Michigan City, Indiana
  - Kentucky Research Group, Louisville, Kentucky
  - Helene Emsellem, MD, Chevy Chase, Maryland
  - Infinity Medical Research, Inc., North Dartmouth, Massachusetts
  - Barrett Clinic, La Vista, Nebraska
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Clinilabs NYC, New York, New York
  - Research Carolina of Huntersville, Huntersville, North Carolina
  - Coastal Carolina Healthcare, New Bern, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Oregon Center for Clinical Investigations,Inc, Salem, Oregon
  - BTC of Lincoln, Lincoln, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Bogan Sleep Consulting, LLC, Columbia, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Tri-State Mountain Neurology, Johnson City, Tennessee
  - Inquest Clinical Research, Baytown, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas
  - Aspen Clinical Research, Orem, Utah
  - Pulmonary Associates of Richmond, Richmond, Virginia
  - Sleep Disorders Centers of the Mid-Atlantic, Vienna, Virginia
  - Swedish Medical Center, Seattle, Washington
- Australia (7):
  - Respiratory Clinical Trials, Adelaide
  - Genesis Sleep Care Queensland, Auchenflower
  - Melbourne Sleep Disorders Centre, East Melbourne
  - The Woolcock Institute of Medical Research, Glebe
  - Royal Melbourne Hospital, Department of Respiratory Medicine, Parkville
  - Gold Coast University Hospital, Respiratory Medicine and Sleep Services, Southport
  - Westmead Hospital, Department of Respiratory and Sleep Medicine, Westmead
- Canada (4):
  - Tri-Hospital Sleep Laboratory West, Mississauga
  - CRIUSMQ- CIUSSSCN, CETS (clinique du sommeil), Québec
  - MedSleep, Toronto
  - Jodha Tishon Inc., Toronto
- Scan Sleep Specialists, Copenhagen, Denmark
- Germany (11):
  - St Hedwig-Krankenhaus, Klinik für Schlaf- und Chronomedizin, Berlin
  - emovis GmbH, Berlin
  - Synexus Berlin Research Centre, Berlin
  - Clinical Trial Center North GmbH & Co. KG, Hamburg
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Klinische Forschung Karlsruhe GmbH, Karlsruhe
  - Studienzentrum Wilhelmshöhe GmbH, Kassel
  - Synexus Leipzig Research Centre, Leipzig
  - Klinikum Rechts der lsar TU München Dept. of Psychiatry and Psychotherapy, München
  - Kinische Forschung Schwerin GmbH, Schwerin
  - ZMS Zentrum für medizinische Studien GmbH, Warendorf
- Italy (4):
  - Ospedale San Raffaele - Centro per i Disturbi del Sonno San Raffaele - Ville-Turro - Pallazzina E, Milan
  - IRCCS FONDAZIONE Istituto Neurologico Nazionale "Casimiro Mondino" - Centro di Ricerca Interdipartimentale per la SSclerosi Multipla (CRISM) -, Pavia
  - Azienda Ospedaliero Universitaria Pisana - Ospedale S. Chiara - Centro di Medicina del Sonno - Clinica Neuroligica - Dipartimento de Neuroscienze, Pisa
  - AOU Citta della Salute e della Scienza - Molinette - SSD Medicina del Sonno, Torino
- Poland (3):
  - PI-House - Centrum Badań Klinicznych, Gdansk
  - Ośrodek Medycyny Study Nurseu Instytutu Psychiatrii i Neurologii (Sleep Disorders Center), Warsaw
  - EMC Instytut Medyczny SA, Przychodnia przy Łowieckiej, Wroclaw
- Serbia (2):
  - General Hospital Bel Medic, Center for Sleep disorders, Belgrade
  - Medigroup - Health Center Dr Ristic (MediGroup Dom zdravlja "Dr Ristic") - Neurology Department, New Belgrade
- Spain (8):
  - Centro Médico Teknon - Medicina del Sueño, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron - Neurophisiology Deparment - Sleep Unit, Barcelona
  - Hospital General de Castellon, Castellon
  - Instituto de Investigaciones del Sueno, Madrid
  - San Carlos University Hospital - Servicio de Neurofisiología Clínica, Madrid
  - Hospital Universitario Araba - Unidad Funcional de Trastornos del Sueño, Vitoria-Gasteiz
  - Hospital MAZ - Neurophisiology and Sleep Department, Zaragoza
- Switzerland (5):
  - KSM Bad Zurzach, Klinik für Schlafmedizin, Bad Zurzach
  - Universitäre Psychiatrische Kliniken Basel (Upk), Basel
  - Universitätsklinik für Neurologie, Inselspital Bern, Schlaf-Wach-Epilepsie-Zentrum, Bern
  - Zentrum für Schlafmedizin Zürcher Oberland, Zürcher RehaZentrum Wald, Wald
  - Zentrum für Schlafmedizin GZO AG Spital Wetzikon, Wetzikon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hudgens S, Phillips-Beyer A, Newton L, Seboek Kinter D, Benes H. Development and Validation of the Insomnia Daytime Symptoms and Impacts Questionnaire (IDSIQ). Patient. 2021 Mar;14(2):249-268. doi: 10.1007/s40271-020-00474-z. Epub 2020 Nov 1. PMID 33131027
- [Result] Mignot E, Mayleben D, Fietze I, Leger D, Zammit G, Bassetti CLA, Pain S, Kinter DS, Roth T; investigators. Safety and efficacy of daridorexant in patients with insomnia disorder: results from two multicentre, randomised, double-blind, placebo-controlled, phase 3 trials. Lancet Neurol. 2022 Feb;21(2):125-139. doi: 10.1016/S1474-4422(21)00436-1. PMID 35065036
- [Derived] Schaedel Z, Bakker TR, Bassetti C, Briasoulis O, Cassel P, Pain S, Palacios S, Palmay C, Silvestri R, Stute P, Tremollieres F, Bertisch SM. Efficacy and safety of daridorexant for the treatment of insomnia disorder in women of menopausal transition age: Insights from a randomized controlled trial. Maturitas. 2025 Dec 23;206:108821. doi: 10.1016/j.maturitas.2025.108821. Online ahead of print. PMID 41506007
- [Derived] Lettieri CJ, Briasoulis O, Leger D, Luyet PP, Pepin JL, Quan SF, Raphelson J, Saskin P, Malhotra A. The Effects of Daridorexant on Patients With Comorbid Insomnia Disorder and Untreated Mild Obstructive Sleep Apnoea: A Post Hoc Subgroup Analysis of a Phase 3, Randomised Clinical Trial. J Sleep Res. 2025 Jul 14:e70135. doi: 10.1111/jsr.70135. Online ahead of print. PMID 40660750
- [Derived] Dauvilliers Y, Braunstein G, Zammit G, Olivieri A, Luyet PP. Effect of daridorexant on nighttime wakefulness and next-morning sleepiness: assessing the transition from night to day in insomnia disorder. Sleep Med. 2025 Jul;131:106523. doi: 10.1016/j.sleep.2025.106523. Epub 2025 Apr 17. PMID 40288253
- [Derived] Di Marco T, Djonlagic I, Dauvilliers Y, Sadeghi K, Little D, Datta AN, Hubbard J, Hajak G, Krystal A, Olivieri A, Parrino L, Puryear CB, Zammit G, Donoghue J, Scammell TE. Effect of daridorexant on sleep architecture in patients with chronic insomnia disorder: a pooled post hoc analysis of two randomized phase 3 clinical studies. Sleep. 2024 Nov 8;47(11):zsae098. doi: 10.1093/sleep/zsae098. PMID 38644625
- [Derived] Phillips-Beyer A, Kawata AK, Kleinman L, Seboek Kinter D, Flamion B. Meaningful Within-Patient Change in Subjective Total Sleep Time in Patients with Insomnia Disorder: An Analysis of the Sleep Diary Questionnaire Using Data from Open-Label and Phase III Clinical Trials. Pharmaceut Med. 2024 Mar;38(2):133-144. doi: 10.1007/s40290-023-00512-9. Epub 2024 Feb 1. PMID 38302765
- [Derived] Citrome L, Juday TR, Lundwall C. Lemborexant and Daridorexant for the Treatment of Insomnia: An Indirect Comparison Using Number Needed to Treat, Number Needed to Harm, and Likelihood to Be Helped or Harmed. J Clin Psychiatry. 2023 Oct 2;84(6):23m14851. doi: 10.4088/JCP.23m14851. PMID 37796657
- [Derived] Dutta S, Singhal S, Shah R, Charan J, Dhingra S, Haque M. Daridorexant as a novel pharmacotherapeutic approach in insomnia: a systematic review and meta-analysis. Expert Opin Drug Saf. 2023 Jul-Dec;22(12):1237-1251. doi: 10.1080/14740338.2023.2243217. Epub 2023 Aug 7. PMID 37526060
- [Derived] Di Marco T, Scammell TE, Meinel M, Seboek Kinter D, Datta AN, Zammit G, Dauvilliers Y. Number, Duration, and Distribution of Wake Bouts in Patients with Insomnia Disorder: Effect of Daridorexant and Zolpidem. CNS Drugs. 2023 Jul;37(7):639-653. doi: 10.1007/s40263-023-01020-9. Epub 2023 Jul 21. PMID 37477771
- [Derived] Phillips-Beyer A, Kawata AK, Kleinman L, Kinter DS. Meaningful Within-Patient Change on the Insomnia Daytime Symptoms and Impacts Questionnaire (IDSIQ): Analysis of Phase III Clinical Trial Data of Daridorexant. Pharmaceut Med. 2023 Jul;37(4):291-303. doi: 10.1007/s40290-023-00484-w. Epub 2023 Jun 7. PMID 37286927
- [Derived] Fietze I, Bassetti CLA, Mayleben DW, Pain S, Seboek Kinter D, McCall WV. Efficacy and Safety of Daridorexant in Older and Younger Adults with Insomnia Disorder: A Secondary Analysis of a Randomised Placebo-Controlled Trial. Drugs Aging. 2022 Oct;39(10):795-810. doi: 10.1007/s40266-022-00977-4. Epub 2022 Sep 13. PMID 36098936
- [Derived] Heidenreich S, Ross M, Chua GN, Seboek Kinter D, Phillips-Beyer A. Preferences of patients for benefits and risks of insomnia medications using data elicited during two phase III clinical trials. Sleep. 2022 Nov 9;45(11):zsac204. doi: 10.1093/sleep/zsac204. PMID 36054921

RESULTS

PARTICIPANT FLOW:
Groups:
- Daridorexant 25 mg; Daridorexant 50 mg: Daridorexant was administered as tablets, orally, once daily in the evening.
- Placebo: Matching placebo was administered as tablets, orally, once daily in the evening.
Period: Overall Study
Arm/Group | Daridorexant 25 mg | Daridorexant 50 mg | Placebo
Started | 310 | 310 | 310
Completed | 288 | 285 | 280
Not Completed | 22 | 25 | 30
Not completed — Death | 1 | 0 | 0
Not completed — Adverse Event | 4 | 2 | 7
Not completed — Other reasons | 3 | 11 | 8
Not completed — Withdrawal by Subject | 13 | 10 | 12
Not completed — Lost to Follow-up | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daridorexant 25 mg | Daridorexant 50 mg | Placebo | Total
Number analyzed (Participants) | 310 | 310 | 310 | 930
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 189 | 189 | 188 | 566
  >=65 years | 121 | 121 | 122 | 364
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (15.3) | 55.5 (15.3) | 55.1 (15.4) | 55.4 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 215 | 199 | 210 | 624
  Male | 95 | 111 | 100 | 306
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 44 | 51 | 146
  Not Hispanic or Latino | 259 | 265 | 259 | 783
  Unknown | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 19 | 30 | 28 | 77
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 1 | 1 | 0 | 2
  Asian | 3 | 4 | 2 | 9
  White | 287 | 274 | 278 | 839
  Other | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 1 in Wake After Sleep Onset (WASO) (Sleep Maintenance)
Description: "Wake After Sleep Onset" is the time spent awake after onset of persistent sleep until lights on, as determined by polysomnography.
Time Frame: From baseline to Month 1 (i.e. for up to 1 month)
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Daridorexant 25 mg | Daridorexant 50 mg | Placebo
Number analyzed (Participants) | 310 | 310 | 310
minutes | -18.40 [-22.126 to -14.674] | -28.98 [-32.668 to -25.299] | -6.20 [-9.928 to -2.475]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in WASO (min) to Month 1 (Daridorexant 25 mg vs placebo); Test type: Other; p < 0.0001, Mixed Models Analysis — Mixed effects model for repeated measures: change from baseline in WASO = baseline WASO + age group (< 65; ≥ 65 years) + treatment + visit + treatment × visit + baseline × visit; LS mean difference to placebo = -12.20, 95% CI 2-sided [-17.435 to -6.961]
Statistical Analysis 2: Comparison: Daridorexant 50 mg vs Placebo; Between-treatment analysis for change from baseline in WASO (min) to Month 1 (Daridorexant 50 mg vs placebo); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS mean difference to placebo = -22.78, 95% CI 2-sided [-27.996 to -17.567]

2. Primary Outcome: Change From Baseline to Month 3 in Wake After Sleep Onset (WASO)
Description: as for outcome 1
Time Frame: From baseline to Month 3 (i.e. for up to 3 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Daridorexant 25 mg | Daridorexant 50 mg | Placebo
Number analyzed (Participants) | 310 | 310 | 310
minutes | -22.97 [-26.955 to -18.988] | -29.41 [-33.399 to -25.427] | -11.11 [-15.131 to -7.088]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in WASO (min) to Month 3 (Daridorexant 25 mg vs placebo); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS mean difference to placebo = -11.86, 95% CI 2-sided [-17.494 to -6.23]
Statistical Analysis 2: Comparison: Daridorexant 50 mg vs Placebo; Between-treatment analysis for change from baseline in WASO (min) to Month 3 (Daridorexant 50 mg vs placebo); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS mean difference to placebo = -18.3, 95% CI 2-sided [-23.945 to -12.661]

3. Primary Outcome: Change From Baseline to Month 1 in Latency to Persistent Sleep (LPS) (Sleep Onset)
Description: "Latency to Persistent Sleep" is the time from start of recording to the beginning of the first continuous 20 epochs (i.e., 10 minutes) scored as non-awake, i.e., epochs scored as either sleep stage 1 (S1), sleep stage 2 (S2), sleep stage 3 (slow wave sleep) or REM, as determined by polysomnography.
Time Frame: From baseline to Month 1 (i.e. for up to 1 month)
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Daridorexant 25 mg | Daridorexant 50 mg | Placebo
Number analyzed (Participants) | 310 | 310 | 310
minutes | -28.17 [-31.509 to -24.827] | -31.20 [-34.506 to -27.896] | -19.85 [-23.177 to -16.515]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in LPS (min) to Month 1 (Daridorexant 25 mg vs placebo); Test type: Other; p = 0.0005, Mixed Models Analysis — Mixed effects model for repeated measures: change from baseline in LPS = baseline LPS + age group (< 65; ≥ 65 years) + treatment + visit + treatment × visit + baseline × visit; LS mean difference to placebo = -8.32, 95% CI 2-sided [-13.014 to -3.629]
Statistical Analysis 2: Comparison: Daridorexant 50 mg vs Placebo; Between-treatment analysis for change from baseline in LPS (min) to Month 1 (Daridorexant 50 mg vs placebo); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference to placebo = -11.35, 95% CI 2-sided [-16.022 to -6.687]

4. Primary Outcome: Change From Baseline to Month 3 in Latency to Persistent Sleep (LPS)
Description: as for outcome 3
Time Frame: From baseline to Month 3 (i.e. for up to 3 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Daridorexant 25 mg | Daridorexant 50 mg | Placebo
Number analyzed (Participants) | 310 | 310 | 310
minutes | -30.73 [-34.037 to -27.417] | -34.80 [-38.118 to -31.490] | -23.13 [-26.464 to -19.803]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in LPS (min) to Month 3 (Daridorexant 25 mg vs placebo); Test type: Other; p = 0.0015, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference to placebo = -7.59, 95% CI 2-sided [-12.265 to -2.923]
Statistical Analysis 2: Comparison: Daridorexant 50 mg vs Placebo; Between-treatment analysis for change from baseline in LPS (min) to Month 3 (Daridorexant 50 mg vs placebo); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference to placebo = -11.67, 95% CI 2-sided [-16.348 to -6.994]

5. Secondary Outcome: Change From Baseline to Month 1 in the Subjective Total Sleep Time (sTST)
Description: "Subjective Total Sleep Time" is the total sleep time reported by the participant in the sleep diary questionnaire. A positive change from baseline indicates an increase in the subjective Total Sleep Time. A negative change from baseline indicates a decrease in subjective Total Sleep Time.
Time Frame: From baseline to Month 1 (i.e. for up to 1 month)
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Daridorexant 25 mg | Daridorexant 50 mg | Placebo
Number analyzed (Participants) | 310 | 310 | 310
minutes | 34.18 [28.718 to 39.645] | 43.62 [38.173 to 49.063] | 21.56 [16.101 to 27.022]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in sTST (min) to Month 1 (Daridorexant 25 mg vs placebo); Test type: Other; p = 0.0013, Mixed Models Analysis — Mixed effects model for repeated measures: change from baseline in sTST = baseline sTST + age group (< 65; ≥ 65 years) + treatment + visit + treatment × visit + baseline × visit; LS mean difference to placebo = 12.62, 95% CI 2-sided [4.953 to 20.288]
Statistical Analysis 2: Comparison: Daridorexant 50 mg vs Placebo; Between-treatment analysis for change from baseline in sTST (min) to Month 1 (Daridorexant 25 mg vs placebo); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; LS mean difference to placebo = 22.06, 95% CI 2-sided [14.405 to 29.708]

6. Secondary Outcome: Change From Baseline to Month 3 in the Subjective Total Sleep Time (sTST)
Description: as for outcome 5
Time Frame: From baseline to Month 3 (i.e. for up to 3 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Daridorexant 25 mg | Daridorexant 50 mg | Placebo
Number analyzed (Participants) | 310 | 310 | 310
minutes | 47.83 [41.333 to 54.328] | 57.67 [51.171 to 64.168] | 37.90 [31.393 to 44.404]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in sTST (min) to Month 3 (Daridorexant 25 mg vs placebo); Test type: Other; p = 0.0334, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; LS mean difference to placebo = 9.93, 95% CI 2-sided [0.782 to 19.082]
Statistical Analysis 2: Comparison: Daridorexant 50 mg vs Placebo; Between-treatment analysis for change from baseline in sTST (min) to Month 3 (Daridorexant 50 mg vs placebo); Test type: Other; p < .00001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; LS mean difference to placebo = 19.77, 95% CI 2-sided [10.623 to 28.918]

7. Secondary Outcome: Change From Baseline to Month 1 in Insomnia Daytime Symptoms and Impacts Questionnaire (IDSIQ) Sleepiness Domain Score
Description: The Insomnia Daytime Symptoms and Impacts Questionnaire (IDSIQ) is a validated patient reported outcome instrument comprising 14 items (each using a numeric rating scale from 0 to 10) grouped into three domains (i.e., sleepiness, mood, and alert/cognition) reflecting daytime impairment of insomnia. The IDSIQ sleepiness domain has 4 items, and the domain score ranges from 0 to a maximum of 40, where a higher score indicates a greater burden. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Time Frame: From baseline to Month 1 (i.e. for up to 1 month)
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Daridorexant 25 mg | Daridorexant 50 mg | Placebo
Number analyzed (Participants) | 310 | 310 | 310
Scores on a scale | -2.77 [-3.316 to -2.225] | -3.77 [-4.309 to -3.224] | -2.02 [-2.566 to -1.476]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in IDSIQ sleepiness domain score to Month 1 (Daridorexant 25 mg vs placebo); Test type: Other; p = 0.0547, Mixed Models Analysis — Mixed effects model for repeated measures: change from baseline in IDSIQ sleepiness domain score = baseline IDSIQ sleepiness domain score + age group (< 65; ≥ 65 years) + treatment + visit + treatment × visit + baseline × visit; LS mean difference to placebo = -0.75, 95% CI 2-sided [-1.515 to 0.015]
Statistical Analysis 2: Comparison: Daridorexant 50 mg vs Placebo; Between-treatment analysis for change from baseline in IDSIQ sleepiness domain score to Month 1 (Daridorexant 50 mg vs placebo); Test type: Other; p < .00001, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; LS mean difference to placebo = -1.75, 95% CI 2-sided [-2.508 to -0.983]

8. Secondary Outcome: Change From Baseline to Month 3 in IDSIQ Sleepiness Domain Score
Description: as for outcome 7
Time Frame: From baseline to Month 3 (i.e. for up to 3 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Daridorexant 25 mg | Daridorexant 50 mg | Placebo
Number analyzed (Participants) | 310 | 310 | 310
Scores on a scale | -4.78 [-5.491 to -4.067] | -5.70 [-6.405 to -4.987] | -3.79 [-4.503 to -3.080]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in IDSIQ sleepiness domain score to Month 3 (Daridorexant 25 mg vs placebo); Test type: Other; p = 0.0534, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; LS mean difference to placebo = -0.99, 95% CI 2-sided [-1.990 to 0.014]
Statistical Analysis 2: Comparison: Daridorexant 50 mg vs Placebo; Between-treatment analysis for change from baseline in IDSIQ sleepiness domain score to Month 3 (Daridorexant 50 mg vs placebo); Test type: Other; p = 0.0002, Mixed Models Analysis; LS mean difference to placebo = -1.90, 95% CI 2-sided [-2.905 to -0.905]

9. Post Hoc Outcome: Change From Baseline to Month 1 in Log-transformed LPS (LSGM Ratio to Baseline)
Description: Post-hoc analyses were performed using log-transformed LPS data, as the LPS values at baseline more closely resembled a log-normal distribution (skewed to the right) than a normal distribution.
Time Frame: From baseline to Month 1 (i.e. for up to 1 month)
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Daridorexant 25 mg | Daridorexant 50 mg | Placebo
Number analyzed (Participants) | 310 | 310 | 310
minutes | 0.49 [0.45 to 0.54] | 0.45 [0.41 to 0.49] | 0.62 [0.57 to 0.67]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in log transformed LPS (min) to Month 1 (Daridorexant 25 mg vs placebo); Test type: Other; p = 0.0003, Mixed Models Analysis — Mixed effects model for repeated measures: log(value/baseline) = log(baseline) + age group(< 65; ≥ 65 years) + treatment + visit + treatment x visit + log(baseline) x visit; LSGM ratio to placebo = 0.79, 95% CI 2-sided [0.70 to 0.90]
Statistical Analysis 2: Comparison: Daridorexant 50 mg vs Placebo; Between-treatment analysis for change from baseline in log transformed LPS (min) to Month 1 (Daridorexant 50 mg vs placebo); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; LSGM ratio to placebo = 0.73, 95% CI 2-sided [0.65 to 0.82]

10. Post Hoc Outcome: Change From Baseline to Month 3 in Log-transformed LPS (LSGM Ratio to Baseline)
Description: as for outcome 9
Time Frame: From baseline to Month 3 (i.e. for up to 3 month)
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Daridorexant 25 mg | Daridorexant 50 mg | Placebo
Number analyzed (Participants) | 310 | 310 | 310
minutes | 0.43 [0.40 to 0.48] | 0.41 [0.37 to 0.45] | 0.56 [0.51 to 0.61]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in log transformed LPS (min) to Month 3 (Daridorexant 25 mg vs placebo); Test type: Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; LSGM ratio to placebo = 0.78, 95% CI 2-sided [0.68 to 0.89]
Statistical Analysis 2: Comparison: Daridorexant 50 mg vs Placebo; Between-treatment analysis for change from baseline in log transformed LPS (min) to Month 3 (Daridorexant 50 mg vs placebo); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; LSGM ratio to placebo = 0.73, 95% CI 2-sided [0.64 to 0.83]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs were AEs that started or worsened on or after the DB study treatment start date up to the earlier of 30 days after DB study treatment end date or the date of enrollment in the ID-078A303 extension study. The planned duration of DB treatment was 84 days ± 2 days, i.e., 12 weeks ± 2 days.
Description: The number of subjects affected is the number of subjects with at least one event.
Arm/Group | Daridorexant 25 mg | Daridorexant 50 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/310 | 0/308 | 0/309
Serious Adverse Events (participants affected / at risk) | 2/310 | 3/308 | 7/309
Other Adverse Events (participants affected / at risk) | 44/310 | 41/308 | 35/309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daridorexant 25 mg (N=310) | Daridorexant 50 mg (N=308) | Placebo (N=309)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daridorexant 25 mg (N=310) | Daridorexant 50 mg (N=308) | Placebo (N=309)
Headache (Nervous system disorders) | 17 (24) | 20 (27) | 12 (18)
Nasopharyngitis (Infections and infestations) | 28 (28) | 24 (26) | 24 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Idorsia for review at least 30 days prior to submission for publication or presentation at a congress. Upon review, Idorsia may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights. Neither the institution nor the investigator should permit publication during such a review period.

DOCUMENTS (2):
  • Study Protocol (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT03545191/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT03545191/SAP_001.pdf